CLINICAL TRIAL: NCT05409820
Title: Comparative Analysis of Hypobaric Versus Hyperbaric Bupivacaine for Spinal Anesthesia in Day-Case Anorectal Surgery: Efficacy, Safety, and Discharge Times
Brief Title: Comparative Analysis of Hypobaric Versus Hyperbaric Bupivacaine for Spinal Anesthesia in Day-Case Anorectal Surgery
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, semih başkan, principle investigator, Ankara City Hospital Bilkent
Other Study IDs: ACH-YALNİZ-001
Record Dates: First submitted 2022-04-17; First posted 2022-06-08 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Anorectal Diseases; Hemorrhoids; Anal Polyp; Pilonidal Sinus; Anal Fissures
Keywords: Day-case Surgery; Spinal Anesthesia; Anorectal Surgery
MeSH Terms: conditions — Rectal Diseases; Hemorrhoids; Pilonidal Sinus; Fissure in Ano

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: use of different spinal anesthesia techniques — Comparison of spinal anesthesia with 5 mg hypobaric bupivacaine and 5 mg hyperbaric bupivacaine in outpatients

SUMMARY:
Spinal anesthesia for anorectal surgery ( fistulotomy, fissure repair, pilonidal sinus excision,hemorrhoidectomy..) is a popular and widely used method characterized by rapid onset, delivery, easy mobilization and short hospital history. In order to minimize complications after spinal anesthesia, the use of lower-dose local anesthesia with the saddle block method has recently become widespread. Bupivacaine is often used for this method. Bupivacaine can be used hypobaric or hyperbaric in spinal anesthesia.

Early mobilization and early discharge are important and necessary in an anorectal disease group that has such a high incidence and does not require rapid surgery and postoperative follow-up and hospitalization.Outpatient surgery is a very suitable surgical procedure for anorectal surgeries.

In the light of all this information, the aim of this study is to evaluate and observe the hemodynamic data, bromage scores, mobilization and discharge of patients who underwent spinal anesthesia with two different techniques.

DETAILED DESCRIPTION:
In this study, it is aimed to reduce long hospital stays and postoperative complications by comparing the postoperative mobilization, urination and discharge times of the patients after spinal anesthesia using 5mg hypobaric and 5 mg hyperbaric bupivacaine in patients who will undergo outpatient anorectal surgery.

After the approval of the ethics committee in the operating room of the Ankara City Hospital, 68 patients who will undergo day surgery due to anorectal disease will be included in the study. This study was planned as observational.

Both genders, American society of anesthesiology(ASA) score 1-2, 68 patients between the ages of 18-65 will be included in the study. The patients will be evaluated in 2 groups of 34 people.

Patients with routine preoperative preparation, ECG, Spo2( oxygen saturation) and non-invasive blood pressure monitoring in the operating room and throughout the study will be included. Written informed consent will be obtained from patients.

ECG, Spo2 and noninvasive blood pressure monitoring of the patients who are taken back to the hospitalization service for postoperative follow-up after the operation will continue. Patients will be followed up with:

half-hourly intervals, first analgesic requirement, urination, mobilization times.

If there are no complications, the patients will be discharged. The next day, patients will be called and questioned in terms of spinal anesthesia-related complications (headache, low back pain, urinary dysfunction…) and their anesthetic satisfaction will be noted.

A total of minimum 68 (n1=34, n2=34) patients with effect size d=0.80, α=0.05 were found to be sufficient for 90% power in the sample size calculation.

Parameters to look at:

Operation time Intraoperative and postoperative vital monitoring need for sedation Time of sensory block to reach s4 dermatome The highest dermatome reached by sensory block Loss time of sensory block Modified bromage scale (5 minutes after spinal cord, end of operation, 1 postoperative 15 minutes, time to zero value) Time to first postoperative analgesic requirement Postoperative urination time Postoperative mobilization time Presence of complications related to spinal anesthesia patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes undergoing anorectal surgery, 18-65 years old, ASA score 1-2 patients

Exclusion Criteria:

* be under the age of 18
* be over 65
* ASA score of 3 and greater than 3
* patients with fever
* those who are pregnant
* Patients with kidney failure
* Patients with hepatic insufficiency
* Patients with heart failure
* Patients with upper respiratory tract symptoms
* Patients with coagulation disorders
* Patients with infection in the lumbar region
* Patients with BMI <18 and BMI >40
* Patients with uncontrolled hypertension, diabetes, pheochromocytoma and thyroid dysfunction
* Those who do not have the ability to read, write or understand the consent form
* Patients who do not want to sign the consent form
* Patients deemed unsuitable by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both sexes undergoing anorectal surgery, 18-65 years old, ASA score 1-2 patients
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Discharge Time | 1 day after surgery
  to determine the time at which patients are ready for discharge

SECONDARY OUTCOMES:
Modified Bromage Scale | 5 minutes after spinal anesthesia End of the surgery (up to 1 hour) Postoperative 15 minutes Postoperative 30 minutes Postoperative 45 minutes Postoperative 60 minutes
  to determine the amount of motor function
Time Of First Analgesic Need | 1 day after surgery
  to measure when the pain started
Urination Time | 1 day after surgery
  to determine the presence of urinary dysfunction
Mobilization Time | 1 day after surgery
  with a modified bromage scale of zero and able to walk unaided
Postoperative Complication | 1 day after surgery
  presence of headache, urinary dysfunction, postoperative nausea and vomiting
Blood Pressure | it is registered in entry, intraop 5.minutes,10.minutes,15.minutes, 20.minutes, 25.minutes, 30.minutes, 35.minutes, 40.minutes, 45.minutes, 50.minutes, 55.minutes,60. minutes ,postoperative 1st hour ,postoperative 2nd hour,postoperative 3rd hour
  systolic, diastolic and mean arterial pressure,to determine the hemodynamic effects of spinal anesthesia
Heart Rate | it is registered in entry, intraop 5.minutes,10.minutes,15.minutes, 20.minutes, 25.minutes, 30.minutes, 35.minutes, 40.minutes, 45.minutes, 50.minutes, 55.minutes,60. minutes ,postoperative 1st hour ,postoperative 2nd hour,postoperative 3rd hour
  to determine the hemodynamic effects of spinal anesthesia
Spo2 | it is registered in entry, intraop 5.minutes,10.minutes,15.minutes, 20.minutes, 25.minutes, 30.minutes, 35.minutes, 40.minutes, 45.minutes, 50.minutes, 55.minutes,60. minutes ,postoperative 1st hour ,postoperative 2nd hour,postoperative 3rd hour
  to determine the hemodynamic effects of spinal anesthesia
Number of Participants with Sedation Need | intraoperative, during surgery
  to determine whether sufficient sensory block has occurred
The Highest Dermatome Reached By The Sensory Block | intraoperative
  to determine whether sufficient sensory block has occurred
S4 Dermatome Sensory Blockage Time | preoperative, intraoperative
  to determine the time it takes for adequate sensory block to occur for surgery
Time to Disappearance of Sensory Block | 1 day after surgery
  to calculate the duration of the effect of spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Semih Başkan, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Honca M, Dereli N, Kose EA, Honca T, Kutuk S, Unal SS, Horasanli E. Low-dose levobupivacaine plus fentanyl combination for spinal anesthesia in anorectal surgery. Braz J Anesthesiol. 2015 Nov-Dec;65(6):461-5. doi: 10.1016/j.bjane.2014.01.007. Epub 2014 Feb 20. PMID 26614142
- [Background] Taspinar V, Sahin A, Donmez NF, Pala Y, Selcuk A, Ozcan M, Dikmen B. Low-dose ropivacaine or levobupivacaine walking spinal anesthesia in ambulatory inguinal herniorrhaphy. J Anesth. 2011 Apr;25(2):219-24. doi: 10.1007/s00540-010-1089-9. Epub 2011 Jan 12. PMID 21225292